CLINICAL TRIAL: NCT03349710
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of Nivolumab or Nivolumab Plus Cisplatin, in Combination With Radiotherapy in Participants With Cisplatin Ineligible and Cisplatin Eligible Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Nivolumab or Nivolumab Plus Cisplatin, in Combination With Radiotherapy in Patients With Cisplatin-ineligible or Eligible Locally Advanced Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9TM; 2017-002676-87 (EudraCT Number)
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Cetuximab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Cohort 1
  Interventions: Biological: Nivolumab; Radiation: Radiotherapy
- Arm B (Experimental): Cohort 1
  Interventions: Drug: Cetuximab; Radiation: Radiotherapy
- Arm C (Experimental): Cohort 2
  Interventions: Biological: Nivolumab; Drug: Cisplatin; Radiation: Radiotherapy
- Arm D (Experimental): Cohort 2
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified day
  Other Names: BMS-936558; Opdivo
  Arms: Arm A; Arm C
Drug: Cetuximab — Specified dose on specified day
  Other Names: Erbitux
  Arms: Arm B
Drug: Cisplatin — Specified dose on specified day
  Arms: Arm C; Arm D
Radiation: Radiotherapy — Specified dose on specified day

SUMMARY:
This study has two, independent, cohorts, both in locally advanced squamous cell head and neck cancer. The purpose of the first cohort is to determine whether nivolumab in combination with radiotherapy is more effective than cetuximab in combination with radiotherapy, in subjects who are ineligible for cisplatin. The purpose of the second cohort is to determine whether nivolumab, cisplatin, and radiotherapy is more effective than cisplatin and radiotherapy in subjects who are eligible to receive cisplatin

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the head and neck (SCCHN) from one of the following primary sites: oral cavity, oropharynx, hypopharynx, and larynx
* Locally advanced disease which is unresectable, or resectable but suitable for an organ sparing approach
* No previous radiotherapy or systemic treatment for SCCHN

Exclusion Criteria:

* Carcinoma originating in the nasopharynx or paranasal sinus, squamous cell carcinoma that originated from the skin and salivary gland or non-squamous histology (e.g., mucosal melanoma), squamous cell carcinoma of unknown primary
* Clinical or radiological evidence of metastatic disease
* Prior radiotherapy that overlaps with radiation fields

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (52):
- United States (21):
  - Pinnacle Research Group, Llc, Anniston, Alabama
  - Cancer Treatment Centers of Phoneix, Goodyear, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCLA Health, Los Angeles, California
  - Cancer Care - Torrance Memorial Physician Network, Redondo Beach, California
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Orlando Health, Inc, Orlando, Florida
  - Winship Cancer Insitute, Emory Crawford Long Hospital, Atlanta, Georgia
  - CTCA Southeastern Region, Newnan, Georgia
  - Lewis Hall Singletary Oncology Center at John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Midwestern Regional medical Center, Zion, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Monter Cancer Center - Center for Advanced Medicine Location, Lake Success, New York
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Upmc- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - The University of Texas MD Anderson Cancer Center-merge, Houston, Texas
  - Inova Health System, Falls Church, Virginia
  - HHP Hematology & Oncology Bremerton, Bremerton, Washington
- France (3):
  - Local Institution, Grenoble
  - Local Institution, Marseille
  - Local Institution, Nice
- Italy (2):
  - Local Institution, Lucca
  - Local Institution, Ravenna
- Japan (12):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Akashi-shi, Hyōgo
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Tsukuba, Ibaraki
  - Local Institution, Isehara, Kanagawa
  - Local Institution, Natori-shi, Miyagi
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Osaka
- Local Institution, Gdynia, Poland
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Yekaterinburg
- South Korea (3):
  - Local Institution, Cheongju-si
  - Local Institution, Jeollanam-do
  - Local Institution, Seoul
- Spain (5):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Majadahonda
  - Local Institution, Valencia
- Taiwan (2):
  - Local Institution, Taichung
  - Local Institution, Tainan
- Local Institution, Izmir, Turkey (Türkiye)

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 Randomized and 73 treated
Groups:
- Arm A (Cohort 1): Nivolumab + Radiotherapy
- Arm B (Cohort 1): Cetuximab + Radiotherapy
- Arm C (Cohort 2): Cisplatin + Nivolumab + Radiotherapy
- Arm D (Cohort 2): Cisplatin + Radiotherapy
Period: Randomized
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Started (= Participants Randomized) | 12 | 10 | 27 | 25
Completed (= Participants Treated) | 12 | 10 | 27 | 24
Not Completed | 0 | 0 | 0 | 1
Period: Treatment Period
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Started (= Participants Treated) | 12 | 10 | 27 | 24
Completed (= Continuing Treatment) | 0 | 0 | 0 | 0
Not Completed | 12 | 10 | 27 | 24
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 2 | 0 | 1
Not completed — Study Drug Toxicity | 1 | 0 | 1 | 1
Not completed — Adverse event unrelated to Study Drug | 2 | 1 | 1 | 1
Not completed — admin reason by sponsor | 0 | 7 | 0 | 19
Not completed — Other Reason | 2 | 0 | 2 | 1
Not completed — completed | 6 | 0 | 18 | 1
Not completed — participant request to discontinue | 0 | 0 | 4 | 0
Not completed — participant withdrew consent | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2) | Total
Number analyzed (Participants) | 12 | 10 | 27 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.5 (8.3) | 74.7 (6.5) | 59.0 (6.6) | 60.8 (7.0) | 64.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 9
  Male | 10 | 8 | 24 | 23 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9 | 2 | 20
  Unknown or Not Reported | 7 | 6 | 18 | 23 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 6 | 15 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 8 | 5 | 16 | 7 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 3 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: Number of Participants with an Adverse Event
Time Frame: 30 Days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants | 12 | 10 | 27 | 24

2. Primary Outcome: Number of Participants With an Serious Adverse Event (SAE)
Description: Number of Participants with an Serious Adverse Event (SAE)
Time Frame: 30 days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants | 5 | 5 | 9 | 6

3. Primary Outcome: Number of Participants With an Adverse Event Leading to Discontinuation
Description: Number of Participants with an Adverse Event Leading to Discontinuation
Time Frame: 30 Days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants | 2 | 3 | 8 | 4

4. Primary Outcome: Number of Participants With an Adverse Event Leading to Dose Modification
Description: Number of Participants with an Adverse Event Leading to dose modification
Time Frame: 30 Days
Population: All Treated Participants
  Dose levels were maintained, no dose modification occurred
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Select Adverse Events
Description: Number of Participants with select adverse events.
  Select Adverse events include: gastrointestinal, hepatic, hypersensitivity/infusion reaction, pulmonary, renal, or skin.
Time Frame: 30 Days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants
  Gastrointestinal | 4 | 3 | 3 | 1
  Hepatic | 1 | 2 | 2 | 3
  Hypersensitivity/Infusion Reaction | 1 | 3 | 0 | 0
  Pulmonary | 0 | 0 | 0 | 0
  Renal | 2 | 1 | 13 | 6
  Skin | 7 | 7 | 12 | 11

6. Primary Outcome: Number of Participants With an Immune-mediated Adverse Event (IMAE)
Description: Number of Participants with an immune-mediated adverse event (IMAE)
Time Frame: 100 days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants
  Non-Endocrine related IMAE | 1 | 0 | 3 | 0
  Endocrine related IMAE | 0 | 0 | 4 | 0

7. Primary Outcome: Time to Onset and Time to Resolution of Immune-related Adverse Events
Description: Time to onset and time to resolution of immune-related adverse events
Time Frame: 100 days
Population: All Treated Participants - Insufficient amount of participants with IMAEs for time to onset and time to resolution
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants Who Experienced Death
Description: Number of Participants who experienced death
Time Frame: 100 days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants | 2 | 2 | 2 | 1

9. Primary Outcome: Number of Participants With an Abnormality in Specific Thyroid Tests
Description: Number of participants with an abnormality in specific thyroid tests
Time Frame: 30 Days
Population: All Treated participants with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 10 | 10 | 27 | 23
Participants
  TSH > ULN | 5 | 1 | 7 | 1
  TSH > ULN WITH TSH <= ULN AT BASELINE | 5 | 1 | 7 | 1
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 4 | 0 | 4 | 0
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 0 | 0 | 2 | 1
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1 | 1 | 1 | 0
  TSH < LLN | 4 | 3 | 16 | 13
  TSH <LLN WITH TSH >= LLN AT BASELINE | 3 | 3 | 13 | 13
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 0 | 9 | 2
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 4 | 1 | 6 | 7
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 2 | 1 | 4

10. Primary Outcome: Number of Participants With an Abnormality in Specific Liver Tests
Description: Number of participants with an abnormality in specific liver tests
Time Frame: 30 days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
Number analyzed (Participants) | 12 | 10 | 27 | 24
Participants
  ALT OR AST > 3XULN | 2 | 0 | 0 | 0
  ALT OR AST> 5XULN | 1 | 0 | 0 | 0
  ALT OR AST> 10XULN | 0 | 0 | 0 | 0
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30DAYS | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 101 days approximately
Arm/Group | Arm A (Cohort 1) | Arm B (Cohort 1) | Arm C (Cohort 2) | Arm D (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 2/12 | 2/10 | 2/27 | 1/24
Serious Adverse Events (participants affected / at risk) | 6/12 | 5/10 | 10/27 | 7/24
Other Adverse Events (participants affected / at risk) | 12/12 | 10/10 | 26/27 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cohort 1) (N=12) | Arm B (Cohort 1) (N=10) | Arm C (Cohort 2) (N=27) | Arm D (Cohort 2) (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Bacillus bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cohort 1) (N=12) | Arm B (Cohort 1) (N=10) | Arm C (Cohort 2) (N=27) | Arm D (Cohort 2) (N=24)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 12 | 8
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 5 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 4 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 6 | 0
Dry eye (Eye disorders) | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 12 | 9
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 6 | 3 | 11 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 17 | 11
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 7 | 6
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Saliva altered (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 4 | 10 | 7
Vomiting (Gastrointestinal disorders) | 1 | 1 | 6 | 8
Asthenia (General disorders) | 2 | 0 | 2 | 2
Fatigue (General disorders) | 4 | 5 | 8 | 3
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 2
Mucosal inflammation (General disorders) | 2 | 2 | 7 | 9
Oedema peripheral (General disorders) | 1 | 0 | 0 | 3
Pain (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 2 | 4 | 2
Xerosis (General disorders) | 0 | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Oral candidiasis (Infections and infestations) | 2 | 1 | 2 | 3
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Incision site inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 4 | 5 | 8 | 12
Recall phenomenon (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 8 | 3
Blood electrolytes abnormal (Investigations) | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 4 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 9 | 8
Platelet count decreased (Investigations) | 0 | 0 | 3 | 1
Protein total decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 3 | 2 | 11 | 7
White blood cell count decreased (Investigations) | 0 | 0 | 7 | 7
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 9 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 5 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 4 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 3
Dysgeusia (Nervous system disorders) | 2 | 2 | 12 | 6
Headache (Nervous system disorders) | 1 | 2 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 3 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 3 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 1
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 7
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 8 | 2
Paranasal sinus hyposecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 8 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 3 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03349710/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03349710/SAP_000.pdf